CLINICAL TRIAL: NCT03995849
Title: Paediatric and Adolescent Radiotherapy Without Anaesthesia Using Audio-Visual Distraction - Are the Patients Moving?
Brief Title: Motion of Kids on Radiation Treatment
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: UHN REB 18-5370
Record Dates: First submitted 2019-06-19; First posted 2019-06-24 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Observational Study
MeSH Terms: interventions — Tomography, Spiral Computed

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Cone Beam CT Scan — In this study, children will receive one CBCT scan before starting RT as part of standard approach. Then after RT, another CBCT scan will be used to measure movement between the beginning and end of RT.

SUMMARY:
At Princess Margaret Cancer Centre, a comprehensive approach to help children stay still during radiation treatment (RT) such as audio-visual distraction (television) is routinely used. These techniques help reduce the need for sedation or general anaesthesia to keep children still to avoid the chance of missing the tumour during RT. This approach has not been systematically evaluated to determine its effectiveness at reducing movement of children receiving RT. The purpose of the study is to measure the movement of children between the beginning and the end of RT to see how much they moved during treatment.

DETAILED DESCRIPTION:
Cone beam CT (CBCT) is a low-dose imaging technique routinely used at Princess Margaret Cancer Centre to check the position of patients before RT. Using CBCT, the doctor is able to reduce the amount of tissues that receive RT because patients can be set-up with greater accuracy to only target the tumour and not harm the surrounding healthy tissue. In this study, children will receive one CBCT scan before starting RT as part of standard approach. Then after RT, another CBCT scan will be used to measure movement between the beginning and end of RT. The information gathered from this study will benefit other patients and cancer centres in the future, who can learn from these methods of using audio-visual distraction so that children have minimal or no motion for a more precise delivery of radiation during cancer treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patient (paediatric or adolescent) age 18 or under receiving RT without anaesthetic or procedural sedation (anaesthetic gas or intravenous sedative medication)

Exclusion Criteria:

* Patients receiving oral midazolam or ketamine are ineligible
* Patient is receiving total body irradiation without CBCT

Max Age: 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Paediatric patients receiving an existing multi-faceted approach to reduce anaesthesia use in paediatric and adolescent radiotherapy (RT)
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2019-10-29 (Actual); Primary Completion 2024-02-05 (Actual); Study Completion 2024-02-05 (Actual)

PRIMARY OUTCOMES:
The proportion of patients that move between pre- and post-RT CBCT acquisitions without anaesthesia. | 12 months
  To determine the proportion of patients with adequate immobilization by measuring motion between pre- and post-RT CBCT acquisitions for patients treated without anaesthesia

SECONDARY OUTCOMES:
Quantitative intra-fraction motion of patients treated with RT without anaesthesia. | 12 months
  To quantitatively determine intra-fraction motion of patients treated with RT without anaesthesia
Factors associated with intra-fraction patient motion. | 12 months
  To evaluate factors associated with intra-fraction patient motion, thus facilitating creation of individualized, patient-specific planning target volumes (PTV)
Perturbations in delivered treatment dose. | 12 months
  To calculate perturbations in delivered treatment dose using dose-accumulation upon on-treatment CBCT images

CONTACTS AND LOCATIONS:
Overall Officials: Derek Tsang, MD, FRCPC, Principal Investigator — Princess Margaret Cancer Centre, University Health Network
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anghelescu DL, Burgoyne LL, Liu W, Hankins GM, Cheng C, Beckham PA, Shearer J, Norris AL, Kun LE, Bikhazi GB. Safe anesthesia for radiotherapy in pediatric oncology: St. Jude Children's Research Hospital Experience, 2004-2006. Int J Radiat Oncol Biol Phys. 2008 Jun 1;71(2):491-7. doi: 10.1016/j.ijrobp.2007.09.044. Epub 2008 Jan 22. PMID 18207663
- [Background] Scott MT, Todd KE, Oakley H, Bradley JA, Rotondo RL, Morris CG, Klein S, Mendenhall NP, Indelicato DJ. Reducing Anesthesia and Health Care Cost Through Utilization of Child Life Specialists in Pediatric Radiation Oncology. Int J Radiat Oncol Biol Phys. 2016 Oct 1;96(2):401-405. doi: 10.1016/j.ijrobp.2016.06.001. Epub 2016 Jun 5. PMID 27475669
- [Background] Khurmi N, Patel P, Koushik S, Daniels T, Kraus M. Anesthesia Practice in Pediatric Radiation Oncology: Mayo Clinic Arizona's Experience 2014-2016. Paediatr Drugs. 2018 Feb;20(1):89-95. doi: 10.1007/s40272-017-0259-8. PMID 28786083
- [Background] Owusu-Agyemang P, Grosshans D, Arunkumar R, Rebello E, Popovich S, Zavala A, Williams C, Ruiz J, Hernandez M, Mahajan A, Porche V. Non-invasive anesthesia for children undergoing proton radiation therapy. Radiother Oncol. 2014 Apr;111(1):30-4. doi: 10.1016/j.radonc.2014.01.016. Epub 2014 Feb 20. PMID 24560754
- [Background] Seiler G, De Vol E, Khafaga Y, Gregory B, Al-Shabanah M, Valmores A, Versteeg D, Ellis B, Mustafa MM, Gray A. Evaluation of the safety and efficacy of repeated sedations for the radiotherapy of young children with cancer: a prospective study of 1033 consecutive sedations. Int J Radiat Oncol Biol Phys. 2001 Mar 1;49(3):771-83. doi: 10.1016/s0360-3016(00)01357-2. PMID 11172961
- [Background] Letourneau D, Wong JW, Oldham M, Gulam M, Watt L, Jaffray DA, Siewerdsen JH, Martinez AA. Cone-beam-CT guided radiation therapy: technical implementation. Radiother Oncol. 2005 Jun;75(3):279-86. doi: 10.1016/j.radonc.2005.03.001. PMID 15890424
- [Background] Guerreiro F, Seravalli E, Janssens GO, van de Ven CP, van den Heuvel-Eibrink MM, Raaymakers BW. Intra- and inter-fraction uncertainties during IGRT for Wilms' tumor. Acta Oncol. 2018 Jul;57(7):941-949. doi: 10.1080/0284186X.2018.1438655. Epub 2018 Feb 19. PMID 29457751
- [Background] Yin FF, Wang Z, Yoo S, Wu QJ, Kirkpatrick J, Larrier N, Meyer J, Willett CG, Marks LB. Integration of cone-beam CT in stereotactic body radiation therapy. Technol Cancer Res Treat. 2008 Apr;7(2):133-9. doi: 10.1177/153303460800700206. PMID 18345702
- [Background] Richmond ND, Pilling KE, Peedell C, Shakespeare D, Walker CP. Positioning accuracy for lung stereotactic body radiotherapy patients determined by on-treatment cone-beam CT imaging. Br J Radiol. 2012 Jun;85(1014):819-23. doi: 10.1259/bjr/54341099. PMID 22665927
- See also: Published Manuscript — https://doi.org/10.1016/j.radonc.2024.110120